CLINICAL TRIAL: NCT07379814
Title: To Investigate the Outcomes of Rectus Abdominis Flap Detrusor Myoplasty for Urinary Retention
Brief Title: Rectus Abdominis Detrusor Myoplasty for Urinary Retention
Acronym: RADM
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Shubham Gupta, Professor, University Hospitals Cleveland Medical Center
Other Study IDs: STUDY20251303
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Urinary Retention; Urinary Retention After Procedure; Urinary Retention Postoperative
Keywords: urinary retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individiuals receiving Rectus Abdominis Detrusor Myoplasty (RADM): Individuals diagnosed with refractory urinary retention that have failed conventional approaches to treat urinary retention such as catheterization and neurostimulation.
  Interventions: Procedure: Rectus Abdominal Detrusor Myoplasty

INTERVENTIONS:
Procedure: Rectus Abdominal Detrusor Myoplasty — In this surgery, the rectus abdominis muscle will be elevated and wrapped circumferentially around the bladder to augment bladder contraction in individuals with bladder acontractility or hypocontractility.

SUMMARY:
This investigates the outcomes of a surgical technique using the patient's own abdominal wall muscles to help contract the bladder in patients with urinary retention

DETAILED DESCRIPTION:
This study is about a surgery called Rectus Abdominis Detrusor Myoplasty (RADM). In this surgery, a small piece of the belly muscle is moved and wrapped around your bladder to help it squeeze and empty urine. Doctors are studying this surgery because current treatments, like catheters or nerve implants, don't always work for people whose bladders don't contract on their own. This study monitors the patients' progress for a year following this surgery.

ELIGIBILITY:
Inclusion Criteria:

* Hypo- or acontractility of the bladder documented on urodynamic testing
* Injury >1 year ago for spinal cord injury patients, no improvement in contractility with time
* Failed sacral nerve stimulation implant for urinary retention treatment (If previously implanted)
* Irreversible non-neurogenic bladder acontractility/hypocontractility (i.e myogenic failure after chronic obstruction, aging, frailty, idiopathic)
* Undergoing RADM

Exclusion Criteria:

* Documented bladder outlet obstruction
* Spinal cord lesion above T12
* Upper motor neuron lesion (i.e. multiple sclerosis, stroke)
* Rectus diastasis, significant abdominal wall hernia, or other anatomic barrier to rectus flap harvest
* Life expectancy <10 years
* Pregnant at time of surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with refractory urinary retention undergoing RADM
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2036-05-01 (Estimated); Study Completion 2036-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Bladder Compliance | 6 Months and 1 Year Post-Op
  Bladder compliance will be calculated as the change in bladder volume divided by the change in detrusor pressure during the filling phase and reported in milliliters per centimeter of water (mL/cm H₂O).
Change in Detrusor Pressure | 6 Months and 1 Year Post-Op
  Detrusor pressure during filling and voiding, including detrusor pressure at maximum flow, will be reported in centimeters of water (cm H₂O).
Change in presence of Detrusor Overactivity | 6 Months and 1 Year Post-Op
  Detrusor overactivity will be recorded as a binary variable (present or absent) based on the occurrence of involuntary detrusor contractions during filling.
Change in Urinary Flow Rate | 6 Months and 1 Year Post-Op
  Maximum urinary flow rate will be reported in milliliters per second (mL/s).
Change In Post-Void Residual Urine Volume in Urine | 6 Months and 1 Year Post-Op
  Post-void residual volume will be measured immediately following voiding and reported in milliliters (mL).

SECONDARY OUTCOMES:
Change in quality of life as measured by the Short-Form 36 (SF-36) | Month 6 and Year 1 Post-Op
  This is a validated questionnaire measuring health-related quality of life through eight domains, covering physical and mental well-being. It's widely used in healthcare to assess overall health perception and functional status. With higher scores indicating greater quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Shubham Gupta, MD, Principal Investigator — University Hospitals Cleveland

IPD SHARING:
Plan to Share IPD: No